CLINICAL TRIAL: NCT04414384
Title: Abdominal Binder and Steps (ABS): A Way to Improve Ambulation Post-Laparotomy in Benign GYN Surgery
Brief Title: Abdominal Binder and Steps Trial
Acronym: ABS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Charles Ascher-Walsh, Associate Professor, Department of Obstetrics, Gynecology, and Reproductive Science, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GCO 19-2072
Record Dates: First submitted 2020-06-01; First posted 2020-06-04 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Post-operative Milestones
Keywords: Post-operative ambulation; Post-operative pain; Abdominal binder; Step counter
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Patients are randomized to either the investigational group (abdominal binder) or control group (no abdominal binder). Those two groups are then both given step counters and their steps are recorded over a two week period.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Abdominal Binder (Experimental): During this time they will wear a step counter and track their steps. This step counter will be returned at the time of their two week visit.
  Interventions: Other: Abdominal Binder; Other: Step Counter
- Control (Other): This group of patients will not wear abdominal binders, but during this time they will wear a step counter and track their steps. This step counter will be returned at the time of their two week visit.
  Interventions: Other: Step Counter

INTERVENTIONS:
Other: Abdominal Binder — Abdominal Binder placement
  Arms: Abdominal Binder
Other: Step Counter — step counter to track steps

SUMMARY:
Large lower abdominal incisions are still used in many types of common gynecologic surgeries. Patients may experience pain and restrictions to ambulation because of this, which can make healing after surgery harder and more complicated. Abdominal binders, through their added abdominal support, may provide a low cost intervention to help people heal. The study team aims to investigate the effects of abdominal binders on walking in the post- gynecologic surgery period.

DETAILED DESCRIPTION:
Laparotomy is a commonly utilized modality for abdominal entry in benign gynecologic surgery despite preference for minimally invasive techniques when surgically feasible. As with other major abdominal surgeries, patients may experience pain and restrictions to ambulation related to the abdominal incision that complicate the postoperative period. Abdominal binders, through their added abdominal support, may provide a low cost, noninvasive intervention to enhance this vital recovery period. Though the use of abdominal binders have been studied extensively in the postcesarean section patient, no report to date exists assessing the effects on abdominal binders in the postoperative course of benign gynecologic surgeries. The study team aims to investigate the effects of abdominal binders on ambulation in the postoperative period after laparotomy for benign gynecologic surgery. The primary outcome is quantitative ambulation via electronic step counter. Secondary outcomes include time to ambulation, quantitative narcotic utilization, visual analogue pain scale, subjective overall wellbeing. With 85% power the study team attempts to calculate a 1200 step difference in means between abdominal binder and control groups using 67 patients per study arm.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Female
* Patients undergoing benign hysterectomy or myomectomy via low-transverse laparotomy.

Exclusion Criteria:

* ASA classification of three or higher
* Malignancy
* Non-English speaking

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2020-06-28 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Daily step counts | Two weeks (until post-operative appointment when step counter is returned)
  Daily step counts taken via electronic step counter over the course of two weeks.

SECONDARY OUTCOMES:
Time to Ambulation | Within 24 hours (post-operative day one)
  Time it takes for patient to begin ambulating post-operatively.
Narcotic utilization | 24-48 hours post-operatively (the typical time from surgery to discharge)
  Quantitative narcotic utilization while inpatient.
Visual analogue pain scale | 24-48 hours post-operatively (the typical time from surgery to discharge)
  Patient's average pain scale as reported to nursing via analogue pain scale. Total scale from 0-10, higher score indicates more pain
Number of participants who thinks there was a benefit | Two weeks (at time of post-operative visit)
  Number of participants who thinks they benefitted from wearing the abdominal binder as reported retrospectively at the two week post-operative visit.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Ascher-Walsh, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Time Frame: Immediately following publication. No end date.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose. To achieve aims in the approved proposal. Email to the primary investigator with IRB-approved proposal.